CLINICAL TRIAL: NCT00854113
Title: A Phase I , Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of EGT0001474 In Healthy Volunteers
Brief Title: Study to Determine the Safety, Tolerability, and Pharmacokinetic (PK) Profile of EGT0001474 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Albert Collinson Ph.D, President and CEO, Theracos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1474-C-328
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Safety and Tolerability of EGT0001474 in Healthy Volunteers
Keywords: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGT0001474 (Experimental): Ascending doses of EGT0001474
  Interventions: Drug: EGT0001474
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EGT0001474 — Oral ascending doses given daily as capsules for up to 14 days
  Other Names: Human SGLT2 inhibitor
  Arms: EGT0001474
Drug: Placebo — Placebo to match EGT0001474
  Other Names: Human SGLT2 inhibitor
  Arms: Placebo

SUMMARY:
This study evaluated the safety, tolerability and pharmacokinetics of single or multiple doses of EGT0001474.

DETAILED DESCRIPTION:
EGT0001474 is an inhibitor of human sodium dependent glucose co-transporter II being developed for the treatment of Type II Diabetes mellitus.

This is a singe center, Phase-1, double blinded,placebo controlled, dose escalation study of single and multiple ascending doses of EGT0001474 in healthy male and female subjects.

In part-1, subjects were randomized to receive single doses of EGT0001474 at 2.5-150 mg or placebo in the ratio of 3:1. In part-2, subjects were randomized to receive 14 daily doses of EGT0001474 at 10, 50 and 150 mg or placebo in the ratio of 4:1. When the various doses were analysed, the maximum dose 150 mg was found to be tolerable. Although there was no serious adverse events, mild adverse events were observed.

This study provided information on human safety, tolerability, PK and pharmacodynamic effects of EGT0001474.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers between the ages of 18 and 55 years inclusive.
* In good health.
* Female subjects must be surgically sterilized or postmenopausal.
* Body mass index (BMI) between 18 kg/m2 and 30 kg/m2 inclusive.
* Non-smoker.
* Negative drug and alcohol screens.

Exclusion Criteria:

* Abnormal ECG
* Sitting blood pressure above 140/90 mmHg on 2 evaluations at least 10 minutes apart at screening
* Treatment with an investigational drug within 30 days or 7 half-lives, whichever is longer.
* Previous treatment with EGT0001474.
* History of drug abuse.
* Febrile illness within 5 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mason W. Freeman, M.D., Study Chair — Massachusetts General Hospital
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 - Single Dose EGT0001474 2.5 mg: Treatment group - received 2.5 mg single dose of EGT0001474
- Part 1 - Single Dose EGT0001474 5 mg: Treatment group- received 5 mg single dose of EGT0001474
- Part 1 -Single Dose EGT0001474 10 mg: Treatment group- received 10 mg single dose of EGT0001474
- Part 1 - Single Dose EGT0001474 25 mg: Treatment group- received 25 mg single dose of EGT0001474
- Part 1 - Single Dose EGT0001474 75 mg: Treatment group- received 75 mg single dose of EGT0001474
- Part 1 - Single Dose EGT0001474 150mg: Treatment group- received 150 mg single dose of EGT0001474
- Part 1 - Single Dose Placebo: Placebo group- received single dose of placebo capsule
- Part 2 - Mutiple Dose EGT0001474 10 mg: Treatment group- received 14 daily doses of EGT0001474 at the dose of 10mg
- Part 2 - Multiple Dose EGT0001474 50 mg: Treatment group-received 14 daily doses of EGT0001474 at the dose of 50mg
- Part 2 - Multiple Dose EGT0001474 150mg: Treatment group-received 14 daily doses of EGT0001474 at the dose of 150mg
- Part 2 - Multiple Dose Placebo: Placebo group- received placebo capsules for 14 days
Period: Overall Study
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 5 | 7 | 8 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6 | 78
Age, Continuous [Mean (Full Range); unit: years] | 43 [29 to 55] | 26 [18 to 31] | 25 [19 to 40] | 32 [18 to 55] | 29 [23 to 35] | 35 [23 to 55] | 33 [19 to 53] | 30 [20 to 44] | 35 [21 to 49] | 22 [18 to 28] | 26 [22 to 32] | 32 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 8 | 6 | 8 | 6 | 30
  Male | 5 | 6 | 6 | 5 | 6 | 6 | 12 | 0 | 2 | 0 | 0 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 12
  Not Hispanic or Latino | 4 | 4 | 5 | 5 | 6 | 6 | 11 | 7 | 5 | 7 | 6 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 3 | 6 | 4 | 6 | 11 | 7 | 5 | 6 | 5 | 64
  White | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 7
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Others | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Pharmacokinetics results. Cmax -Maximum plasma drug concentration
Time Frame: Part-1 (Single dose) measured in 1 day and part 2 (multiple doses) measured in 14 days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6
ng/ml | 12.7 (1.08) | 28 (10.2) | 90.7 (31.7) | 194 (53.3) | 537 (198) | 1183 (434) | NA (NA) — Placebo did not receive EGT001474 drug. | 85.7 (27.9) | 465 (126) | 1202 (345) | NA (NA) — Placebo did not receive EGT001474 drug.

2. Primary Outcome: Tmax
Description: Pharmacokinetics results. Time to maximum plasma drug concentration (Tmax) was calculated for each groups
Time Frame: Part-1 (Single dose) measured in 1 day and part 2 (multiple doses) measured in 14 days
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6
hour | 4 [4 to 6] | 2.01 [1 to 4] | 2 [1 to 4] | 1.51 [1 to 6] | 1.5 [1 to 3] | 1.5 [1 to 4] | NA [NA to NA] — Placebo did not receive EGT001474 drug | 2.01 [1 to 6] | 1 [1 to 6.05] | 1 [1 to 1] | NA [NA to NA] — Placebo did not receive EGT001474 drug

3. Primary Outcome: AUC 0-t
Description: Pharmacokinetics results. AUC 0-t - Are under plasma concentration-time curve from time 0 time t.
Time Frame: Part-1 (Single dose) measured in 1 day and part 2 (multiple doses) measured in 14 days
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6
ng*hr/ml | 67.4 (13.9) | 126 (33.8) | 388 (108) | 1200 (320) | 2564 (607) | 6412 (1179) | NA (NA) — Placebo did not receive EGT001474 drug. | 432 (89.5) | 2146 (539) | 7733 (1957) | NA (NA) — Placebo did not receive EGT001474 drug.

4. Primary Outcome: t1/2
Description: Pharmacokinetics results.t 1/2 - apparent terminal half life
Time Frame: Part-1 (Single dose) measured in 1 day and part 2 (multiple doses) measured in 14 days
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6
hour | 3.66 (0.559) | 4.19 (1.3) | 5.81 (1.38) | 9.71 (3.28) | 9.27 (1.60) | 11.4 (2.49) | NA (NA) — Placebo did not receive EGT001474 drug. | 9.03 (1.44) | 9.02 (2.38) | 10.3 (1.98) | NA (NA) — Placebo did not receive EGT001474 drug.

5. Primary Outcome: AUC 0 -24
Description: Pharmacokinetics results. Area under the plasma concentration-time curve from time 0 to 24 hours post-dose.
Time Frame: Part-1 (Single dose) measured in 1 day and part 2 (multiple doses) measured in 14 days
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6
ng*hr/ml | 85.6 (9.67) | 145 (34.4) | 392 (99.8) | 1121 (264) | 2383 (527) | 5828 (1080) | NA (NA) — Placebo did not receive EGT001474 drug. | 412 (73.8) | 1983 (443) | 6939 (1675) | NA (NA) — Placebo did not receive EGT001474 drug.

6. Primary Outcome: Terminal Rate Constant.
Description: Pharmacokinetics results. Terminal rate constant was estimated by linear regression of logarithmic transformed concentration versus time data
Time Frame: Part-1 (Single dose) measured in 1 day and part 2 (multiple doses) measured in 14 days
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6
L/hr | 0.193 (0.0314) | 0.177 (0.0456) | 0.126 (0.0373) | 0.0799 (0.0308) | 0.0765 (0.0117) | 0.0637 (0.0158) | NA (NA) — Placebo did not receive EGT001474 drug. | 0.0783 (0.0117) | 0.0818 (0.023) | 0.0697 (0.0143) | NA (NA) — Placebo did not receive EGT001474 drug.

7. Primary Outcome: CL/F
Description: Pharmacokinetics results. Apparent oral clearance
Time Frame: Part-1 (Single dose) measured in 1 day and part 2 (multiple doses) measured in 14 days
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6
L/hr | 28.9 (2.89) | 35.3 (8.24) | 25.9 (7.59) | 21.2 (5.18) | 30.1 (8.51) | 23.1 (3.67) | NA (NA) — Placebo did not receive EGT001474 drug. | 24.9 (4.45) | 26.4 (6.49) | 22.6 (4.67) | NA (NA) — Placebo did not receive EGT001474 drug.

8. Primary Outcome: VZ/F
Description: Pharmacokinetic results. Apparent volume of distribution
Time Frame: Part-1 (Single dose) measured in 1 day and part 2 (multiple doses) measured in 14 days
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 8 | 8 | 6
Liters | 154 (37.1) | 222 (121) | 208 (49.5) | 287 (105) | 398 (109) | 385 (121) | NA (NA) — Placebo did not receive EGT001474 drug. | 319 (39.3) | 327 (54.2) | 333 (84.2) | NA (NA) — Placebo did not receive EGT001474 drug.

ADVERSE EVENTS:
Arm/Group | Part 1 - Single Dose EGT0001474 2.5 mg | Part 1 - Single Dose EGT0001474 5 mg | Part 1 -Single Dose EGT0001474 10 mg | Part 1 - Single Dose EGT0001474 25 mg | Part 1 - Single Dose EGT0001474 75 mg | Part 1 - Single Dose EGT0001474 150mg | Part 1 - Single Dose Placebo | Part 2 - Mutiple Dose EGT0001474 10 mg | Part 2 - Multiple Dose EGT0001474 50 mg | Part 2 - Multiple Dose EGT0001474 150mg | Part 2 - Multiple Dose Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/8 | 0/8 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 3/6 | 3/6 | 3/6 | 3/6 | 3/6 | 3/12 | 5/8 | 6/8 | 7/8 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - Single Dose EGT0001474 2.5 mg (N=6) | Part 1 - Single Dose EGT0001474 5 mg (N=6) | Part 1 -Single Dose EGT0001474 10 mg (N=6) | Part 1 - Single Dose EGT0001474 25 mg (N=6) | Part 1 - Single Dose EGT0001474 75 mg (N=6) | Part 1 - Single Dose EGT0001474 150mg (N=6) | Part 1 - Single Dose Placebo (N=12) | Part 2 - Mutiple Dose EGT0001474 10 mg (N=8) | Part 2 - Multiple Dose EGT0001474 50 mg (N=8) | Part 2 - Multiple Dose EGT0001474 150mg (N=8) | Part 2 - Multiple Dose Placebo (N=6)
Application Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1) — General disorders and administrative site conditions
Application Site Irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General disorders and administrative site conditions
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General disorders and administrative site conditions
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General disorders and administrative site conditions
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General disorders and administrative site conditions
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — General disorders and administrative site conditions
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Head Discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharangeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes